CLINICAL TRIAL: NCT00933166
Title: Assessing the Performance of Lotrafilcon A Lenses During a Three Month Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-335-C-014v2
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lotrafilcon A (Experimental): Investigational contact lens worn in both eyes for three months
  Interventions: Device: Lotrafilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon A contact lens — Investigational silicone hydrogel, single vision, soft contact lens worn on a daily wear basis, flexible wear basis, or extended wear basis for three months

SUMMARY:
The purpose of this trial is to assess the performance of an investigational contact lens over a three month period.

ELIGIBILITY:
Inclusion Criteria:

* On examination, have ocular findings considered to be "normal," and which would not prevent a participant from safely wearing contact lenses.
* Be willing and able to follow instructions and meet the schedule of follow-up visits as defined in the informed consent.
* Be able to wear the study lenses in the available powers.
* Currently wear contact lenses for a minimum of 5 days a week, and at least 8 hours a day.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks of enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in an ophthalmic clinical trial.
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* History of corneal refractive surgery.
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lotrafilcon A
Started | 169
Completed | 151
Not Completed | 18
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 9
Not completed — Unavailable | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 169
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Comfort After Insertion
Description: Comfort after insertion (30 seconds to 1 minute) as interpreted and reported by the participant on a questionnaire as a single, retrospective evaluation of three months' wear time. Comfort after insertion was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 3 months
Population: Analysis was per protocol and excluded ten major protocol deviations as determined by masked review. Eighteen participants discontinued prior to the Month 3 visit. Nineteen participants responded N/A due to reasons such as continual wear.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 122
Units on a Scale | 9.0 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 4 months, 16 days.
Arm/Group | Lotrafilcon A
Serious Adverse Events (participants affected / at risk) | 0/169
Other Adverse Events (participants affected / at risk) | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.